CLINICAL TRIAL: NCT03248622
Title: Hepatitis B Reactivation During Treatment With Direct-Acting Antiviral Agents for Chronic Hepatitis C Infection
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999917099; 17-DK-N099
Record Dates: First submitted 2017-08-11; First posted 2017-08-14 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Hepatitis B
Keywords: Incidence; Hepatitis B Surface Antigen; Decompensation
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Anti-HBc positive: Anti-HBc positive
- HCV positive Cohort: HCV positive Cohort

SUMMARY:
Background:

Treatment of some diseases can suppress the immune system. This can cause other conditions to reactivate. Recent cases have shown that hepatitis B virus (HBV) reactivates in people who had already recovered from it during treatment for chronic hepatitis C (CHC). Their treatment was direct-acting antiviral (DAA) agents. Researchers want to see how common this reactivation is. They want to learn what the effects are. They will study data that have already been collected.

Objectives:

To study HBV reactivation in people with CHC and resolved HBV infection who are being treated with interferon-free DAA-based therapy.

Eligibility:

Data were collected from adults 18 and older in studies that were done in 2012 and 2016.

Design:

Researchers will screen the records from the previous studies. They will identify participants who had HBV infection before they got DAA-based treatment.

Researchers will take data from those records. This will include data on:

* Age, sex, race, and ethnicity
* Treatment and disease status
* Lab results

Researchers will test stored samples. They will test samples that were taken before, during, and after treatment. They will check if HBV was reactivated. They will also check if other clinical outcomes occurred.

DETAILED DESCRIPTION:
Reactivation of hepatitis B is well known to occur with immunosuppression as in the setting of high dose immunosuppressive therapy, cancer chemotherapy and bone marrow or stem cell transplantation. It is usually subclinical but at times can manifest as an acute hepatitis, hepatic decompensation and death. Often times this leads to interruption of cancer chemotherapy.

Recently, several case reports and case series have revealed evidence of hepatitis B virus (HBV) reactivation in previously recovered persons being treated for chronic hepatitis C (CHC) with direct-acting antiviral (DAA) agents. Given the severity of some cases, the U.S. Food and Drug Administration (FDA) has issued a Black Box warning regarding the risk of HBV reactivation to HCV DAA labeling to screen all hepatitis C patients for HBV before initiation of therapy and to monitor those with previous HBV infection for signs of reactivation while on treatment. However, since the FDA warning, retrospective experiences on clinical trials have failed to reveal evidence of viral reactivation. Further, the frequency of HBV reactivation and its risk factors and monitoring frequency in HCV patients receiving Interferon-free DAA therapy are yet unknown. Hence, we aim to conduct a multicenter retrospective analysis to investigate these issues.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Adult patients (greater than or equal to 18 years) with CHC who underwent treatment with an Interferon-free DAA-based therapy.
* Evidence of resolved HBV infection prior to starting interferon-free DAAbased therapy (HBsAg-negative with positive anti-HBc +/- positive anti-HBs)

EXCLUSION CRITERIA:

- Treatment with Nucleos(t)ide Analogues (NA) active against HBV prior to initiation of interferon-free DAA therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hepatitis C who were anti-HBc positive and who received treatment with a direct acting antiviral agent.
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2017-06-03 (Actual); Primary Completion 2019-05-28 (Actual); Study Completion 2019-05-28 (Actual)

PRIMARY OUTCOMES:
The rate of HBV reactivation among patient with resolved HBV infection undergoing Interferon-free DAA-based therapy for HCV infection. | From initiation of treatment to 24 weeks post-treatment
  Detection of HBV DNA or HBsAg and elevated ALT level

CONTACTS AND LOCATIONS:
Overall Officials: Marc G Ghany, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institute of Diabetes and Digestive and Kidney Disorders (NIDDK), Bethesda, Maryland, United States